CLINICAL TRIAL: NCT04252950
Title: Community-based Exercise to Improve Physical Functioning and Cardiovascular Health Following Revascularization for Peripheral Artery Disease
Brief Title: Community-based Exercise Following Revascularization for PAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SON-2020-28532
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Artery Disease
Keywords: PAD; peripheral artery disease; claudication; revascularization; community-based exercise
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CB-SET Treatment (Experimental): Participants randomized to this group will receive a community-based structured exercise therapy (CB-SET) along with the standard of care (revascularization)
  Interventions: Behavioral: CB-SET; Procedure: Revascularization
- Control (Active Comparator): Participants randomized to this group will receive standard of care (revascularization)
  Interventions: Procedure: Revascularization

INTERVENTIONS:
Behavioral: CB-SET — Community-based structured exercise therapy (CB-SET) programs for PAD have potential merit as an alternative to hospital-based SET, as they may provide similar benefit to hospital-based programs but in a convenient location for the exercise to be completed
  Arms: CB-SET Treatment
Procedure: Revascularization — Endovascular revascularization is a primary treatment option for patients with PAD

SUMMARY:
The primary goal of this clinical trial is to evaluate whether a community-based structured exercise therapy (CB-SET) intervention, which could be accessible and easily disseminated, adds benefit to peripheral artery disease (PAD) patients undergoing revascularization (REVASC) to improve their function and cardiovascular health.

DETAILED DESCRIPTION:
Training (T): Patients assigned to the control group will receive verbal advice to exercise but will receive no other training following their revascularization and outcome assessments. Patients in the intervention group will receive supervised SET in the exercise physiology laboratory for one week (3 sessions) following their REVASC and outcome assessments. Patients will then receive 11 weeks of community-based structured exercise therapy (CB-SET) with training, monitoring, and coaching (TMC) and public health elements at home or in the place of their choosing. Patients will be visited by study staff where walking exercise will take place (1 visit per month, 3 total community visits). The purpose of the initial supervised SET is to educate patients about how to exercise and to address any questions they may have (part of the training component of TMC).

Monitoring (M): Participants will be monitored with a piezoelectric accelerometer over the duration of the 12 total weeks to determine total volume of activity. Participants in both groups will be asked to wear the monitors continuously for 7 days per week over a 10 hour period for each day. This amount of activity monitoring has been successfully used in previous studies (minimal user burden, low profile devices). Additionally, participants in both groups will be reminded to wear the monitor during any walking sessions they perform with intent of exercise. The investigators will determine exercise compliance separately for both groups, and participants in the intervention group will be asked to record details about the CB-SET sessions in a provided exercise log (as conducted in a pilot studies). Data from the piezoelectric accelerometers, which are capable of collecting and storing data for ~6 weeks, will be downloaded and reset at the community visits (1 per month). Control participants will be mailed a new device every 4 weeks (with pre-paid mailers given to control participants for return and subsequent download by staff) or will exchange the device during optional once per month visits to the exercise laboratory. At these visits, control pariticipants will have resting heart rate and blood pressure assessed but no CB-SET program will be applied to ensure these participants receive the standard of care regarding home exercise (upfront advice to walk). Participants in the intervention group will also be given commercially available piezoelectric hip pedometers (Omron), which have an interface to track steps, to monitor their own activity. Weekly phone calls (telehealth) will be conducted by study staff with specific prompting to gain a better evaluation of how much and how often intervention group participants are walking (a feasible process evaluation used in the preliminary studies). Questions included to assist in determining treatment fidelity (ensuring the intervention is delivered as intended) during phone calls and from the exercise log: 1) date and start/end times of walking exercise for each session, 2) number of rest stops needed while walking (and reasons for stopping), 3) questions regarding usage of the piezoelectric accelerometer (instructions for use given to participants), 4) number of steps measured from the hip pedometer, 5) what route the participant chose to use for walking as initially defined by the environmental audit (see section below for more details), and 6) what barriers or facilitators the participant encountered during the session ("Any problems while walking around your neighborhood?"). Additionally, participants will be strongly encouraged to walk with family, friends, and pets to increase walking activity. Participants in both groups will receive a smartphone with an application called Daynamica, which will allow users to indicate and store the location where they complete their community-based activities and to annotate specific exercise sessions or other physical activity episodes. Participants in the control group will receive monthly phone calls only to assess the occurrence of any adverse events and to schedule the optional in-hospital visit.

Coaching (C): The investigators will employ an operational coaching model that will provide training guidance and help addressing local barriers to exercise training in the community setting as well as promoting or reinforcing facilitators for each individual participant in the CB-SET intervention group. This will include: 1) educational print materials and 2) environmental auditing. Educational materials developed by Vascular Cures will include informational outreach activities that have been cited as strategies to promote walking by the Task Force Community Preventive Services. Additionally, in providing control participants with the accelerometers, the investigators are in essence providing them "attention", in addition to the monthly phone calls and optional in-hospital "check-ups" with controls. This attention-control design is meant to provide definitive findings that the substantive aspects of the CB-SET program are efficacious and not the result of simply increased contact time with intervention group participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving Revascularization for aorto-iliac and/or femoral-popliteal disease in at least one limb
* Patients with focal and/or diffuse peripheral artery disease
* Bilateral Revascularization patients will also be included
* Ability to participate in an exercise program

Exclusion Criteria:

* Lower extremity amputation(s) which interfere(s) with walking on the treadmill
* Individuals with critical limb ischemia defined by ischemic rest pain or ischemic ulcers/gangrene on the lower extremities
* PAD of non-atherosclerotic nature (e.g., fibromuscular dysplasia, irradiation, endofibrosis).
* Coronary artery bypass grafts or major surgical procedures within 6 months prior to screening
* Individuals whose walking exercise is primarily limited by symptoms of chronic obstructive pulmonary disease, angina, or heart failure
* Individuals who have had a myocardial infarction within 3 months prior to screening
* Individuals who have had a transient ischemic attack or stroke 3 months prior to screening
* Individuals with uncontrolled hypertension (≥180 systolic or ≥100 diastolic resting blood pressure) during screening
* Treatment with pentoxifylline or cilostazol for the treatment of claudication 4 weeks prior to screening. Patients can be reconsidered for study inclusion following a 1-month washout period
* Poorly controlled diabetes defined as glycated hemoglobin >12%
* Abnormal results of blood work not conducive to safely participate in an exercise trial (e.g., anemic, electrolyte abnormalities)
* Inability to speak English
* Other clinically significant cardiovascular, pulmonary, renal, endocrine, hepatic, neurological, psychiatric, immunological, gastrointestinal, hematological, or metabolic disease that is, in the opinion of the study team, not stabilized or may otherwise confound the results of the study

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Peak Walking Time (PWT) | Baseline, 12 weeks
  Participants will perform graded exercise tests conducted on a treadmill with continuous electrocardiogram monitoring. Participants will run at a constant speed of 2.0 miles/hour, starting at 0% grade. Every 2 min the grade is increased 2% until maximal claudication limits exercise.
  PWT (reported in minutes) will be recorded as the maximal time a participant can walk on the treadmill before having to stop due to severe claudication (assessed using the Claudication Symptom Rating Scale which ranges from 1-5 with 1=no pain, 2=onset claudication, 3=mild, 4=moderate, and 5=severe).

SECONDARY OUTCOMES:
Change in Claudication Onset Time (COT) | Baseline, 12 weeks
  Participants will perform graded exercise tests conducted on a treadmill with continuous electrocardiogram monitoring. Participants will run at a constant speed of 2.0 miles/hour, starting at 0% grade. Every 2 min the grade is increased 2% until maximal claudication limits exercise.
  COT (reported in minutes) will be obtained with the patient pointing to the pain scale at the initial presentation of leg pain (assessed using the Claudication Symptom Rating Scale which ranges from 1-5 with 1=no pain, 2=onset claudication, 3=mild, 4=moderate, and 5=severe).
Change in VO2max | Baseline, 12 weeks
  VO2 max is the maximum rate of oxygen consumption measured during incremental exercise. Participants will perform graded exercise tests conducted on a treadmill while oxygen consumption is measured and recorded. Maximum rate of oxygen consumption during exercise will be reported in mL/kg*min-1.
Total Volume of Exercise | 12 weeks
  Patients will be monitored with a piezoelectric accelerometer over the duration of the 12 total weeks to determine total volume of activity. The average minutes of activity per day will be reported.
Adherence to Exercise | 12 weeks
  Participants will be given a StepWatch accelerometer. Exercise compliance will be calculated for PAD participants as the total number of completed sessions divided by 36 (3 sessions/week for 12 weeks).
Change in Walking Impairment Questionnaire (WIQ) Distance Subcategory | Baseline, 12 weeks
  In the Walking Impairment Questionnaire distance subcategory, participants are asked to rate the degree of difficulty walking specific distances on a scale from 0 to 4. A score of 0 indicates the inability to walk the distance specified by the question while a score of 4 represents no difficulty. The graded sub-score is multiplied by a pre-specified weight for each sub-category: distance, speed, and number of flights of stairs. The products of these subscores are summed and divided by the maximum possible score to obtain a percent score, ranging from 0 (inability to perform item) to 100 (no difficulty in performing item).
Change in Walking Impairment Questionnaire (WIQ) Speed Subcategory | Baseline, 12 weeks
  In the Walking Impairment Questionnaire speed subcategory, participants are asked to rate the degree of difficulty walking one block at specific speeds, ranging from walking slowly to jogging, on a scale from 0 to 4. A score of 0 indicates the inability to walk the distance specified by the question while a score of 4 represents no difficulty. The graded sub-score is multiplied by a pre-specified weight for each sub-category: distance, speed, and number of flights of stairs. The products of these subscores are summed and divided by the maximum possible score to obtain a percent score, ranging from 0 (inability to perform item) to 100 (no difficulty in performing item).
Change in Walking Impairment Questionnaire (WIQ) Stair-Climbing Subcategory | Baseline, 12 weeks
  In the Walking Impairment Questionnaire stair-climbing subcategory, participants are asked to rate the degree of difficulty climbing a specified number of stair flights, ranging from 1 to 3 stair flights, on a graded scale of 0 to 4. A score of 0 indicates the inability to climb the flights specified by the question while a score of 4 represents no difficulty. The graded sub-score is multiplied by a pre-specified weight for each sub-category: distance, speed, and number of flights of stairs. The products of these subscores are summed and divided by the maximum possible score to obtain a percent score, ranging from 0 (inability to perform item) to 100 (no difficulty in performing item).
Change in SF-36 Physical Component Summary | Baseline, 12 weeks
  The SF-36 has eight scaled subscores (Vitality, Physical functioning, Bodily pain, General health perceptions, Physical role functioning, Emotional role functioning, Social role functioning, Mental health). These subscores are weighted sums of the questions in each section. Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability.
Change in SF-36 Mental Component Summary | Baseline, 12 weeks
  The SF-36 has eight scaled subscores (Vitality, Physical functioning, Bodily pain, General health perceptions, Physical role functioning, Emotional role functioning, Social role functioning, Mental health). These subscores are weighted sums of the questions in each section. Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability.
Change in PADQOL Factor 1: Social Relationships and Interactions | Baseline, 12 weeks
  The Peripheral Artery Disease Quality of Life (PADQOL) is a 38-item survey assessing 5 quality of life factors of PAD patients: Social relationships and interactions; Self-concept and feelings; Symptoms and limitations in physical functioning; Fear and uncertainty; and Positive adaptation. Items are scored on a scale of 1 (strongly agree) to 6 (strongly disagree). 5 factor scores are calculated by summing all items in that factor. These factor scores are labeled F1- F5. The factor totals are then transformed into percentiles using the formula: [(sum of scores on factor items - # of factor items) / (5 * # of factor items)]*100 = factor percentile. Total factor scores range from 0 to 100 with higher scores indicating greater quality of life.
Change in PADQOL Factor 2: Self-concept and Feelings | Baseline, 12 weeks
  The Peripheral Artery Disease Quality of Life (PADQOL) is a 38-item survey assessing 5 quality of life factors of PAD patients: Social relationships and interactions; Self-concept and feelings; Symptoms and limitations in physical functioning; Fear and uncertainty; and Positive adaptation. Items are scored on a scale of 1 (strongly agree) to 6 (strongly disagree). 5 factor scores are calculated by summing all items in that factor. These factor scores are labeled F1- F5. The factor totals are then transformed into percentiles using the formula: [(sum of scores on factor items - # of factor items) / (5 * # of factor items)]*100 = factor percentile. Total factor scores range from 0 to 100 with higher scores indicating greater quality of life.
Change in PADQOL Factor 3: Symptoms and Limitations in Physical Functioning | Baseline, 12 weeks
  The Peripheral Artery Disease Quality of Life (PADQOL) is a 38-item survey assessing 5 quality of life factors of PAD patients: Social relationships and interactions; Self-concept and feelings; Symptoms and limitations in physical functioning; Fear and uncertainty; and Positive adaptation. Items are scored on a scale of 1 (strongly agree) to 6 (strongly disagree). 5 factor scores are calculated by summing all items in that factor. These factor scores are labeled F1- F5. The factor totals are then transformed into percentiles using the formula: [(sum of scores on factor items - # of factor items) / (5 * # of factor items)]*100 = factor percentile. Total factor scores range from 0 to 100 with higher scores indicating greater quality of life.
Change in PADQOL Factor 4: Fear and Uncertainty | Baseline, 12 weeks
  The Peripheral Artery Disease Quality of Life (PADQOL) is a 38-item survey assessing 5 quality of life factors of PAD patients: Social relationships and interactions; Self-concept and feelings; Symptoms and limitations in physical functioning; Fear and uncertainty; and Positive adaptation. Items are scored on a scale of 1 (strongly agree) to 6 (strongly disagree). 5 factor scores are calculated by summing all items in that factor. These factor scores are labeled F1- F5. The factor totals are then transformed into percentiles using the formula: [(sum of scores on factor items - # of factor items) / (5 * # of factor items)]*100 = factor percentile. Total factor scores range from 0 to 100 with higher scores indicating greater quality of life.
Change in PADQOL Factor 5: Positive Adaptation | Baseline, 12 weeks
  The Peripheral Artery Disease Quality of Life (PADQOL) is a 38-item survey assessing 5 quality of life factors of PAD patients: Social relationships and interactions; Self-concept and feelings; Symptoms and limitations in physical functioning; Fear and uncertainty; and Positive adaptation. Items are scored on a scale of 1 (strongly agree) to 6 (strongly disagree). 5 factor scores are calculated by summing all items in that factor. These factor scores are labeled F1- F5. The factor totals are then transformed into percentiles using the formula: [(sum of scores on factor items - # of factor items) / (5 * # of factor items)]*100 = factor percentile. Total factor scores range from 0 to 100 with higher scores indicating greater quality of life.
Change in PADQOL Question 21: Job/Work | Baseline, 12 weeks
  The Peripheral Artery Disease Quality of Life (PADQOL) is a 38-item survey assessing 5 quality of life factors of PAD patients: Social relationships and interactions; Self-concept and feelings; Symptoms and limitations in physical functioning; Fear and uncertainty; and Positive adaptation. Items are scored on a scale of 1 (strongly agree) to 6 (strongly disagree). 5 factor scores are calculated. 3 items (Q21, Q23, and Q24) are not included in any of the factors but are instead reported individually. The raw score of question 21 is transformed using the following formula: [(Q21 - 1) / 5] * 100 = JOB percentile. Final scores range from 0 to 100 with higher scores indicating better quality of life.
Change in PADQOL Question 23: Sex | Baseline, 12 weeks
  The Peripheral Artery Disease Quality of Life (PADQOL) is a 38-item survey assessing 5 quality of life factors of PAD patients: Social relationships and interactions; Self-concept and feelings; Symptoms and limitations in physical functioning; Fear and uncertainty; and Positive adaptation. Items are scored on a scale of 1 (strongly agree) to 6 (strongly disagree). 5 factor scores are calculated. 3 items (Q21, Q23, and Q24) are not included in any of the factors but are instead reported individually. The raw score of question 23 is reserve scored and then transformed using the following formula: [(RQ23 - 1) / 5] * 100 = SEX percentile. Final scores range from 0 to 100 with higher scores indicating better quality of life.
Change in PADQOL Question 24: Intimate Relationships | Baseline, 12 weeks
  The Peripheral Artery Disease Quality of Life (PADQOL) is a 38-item survey assessing 5 quality of life factors of PAD patients: Social relationships and interactions; Self-concept and feelings; Symptoms and limitations in physical functioning; Fear and uncertainty; and Positive adaptation. Items are scored on a scale of 1 (strongly agree) to 6 (strongly disagree). 5 factor scores are calculated. 3 items (Q21, Q23, and Q24) are not included in any of the factors but are instead reported individually. The raw score of question 24 is reserve scored and then transformed using the following formula: [(RQ24 - 1) / 5] * 100 = IR percentile. Final scores range from 0 to 100 with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Mays, PhD, MPH, MS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States